CLINICAL TRIAL: NCT03281213
Title: No Impact of Gender on Acute Postthoracotomy Pain - a Retrospective Analysis
Brief Title: Acute Postthoracotomy Pain - Impact of Gender
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Auinger, Daniel MD, Dr. med. univ., Medical University of Graz
Other Study IDs: genderthorpain
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Gender; Postoperative Pain; Thoracotomy; Analgesia
MeSH Terms: conditions — Coitus; Pain, Postoperative; Agnosia | interventions — Thoracotomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female
  Interventions: Other: Thoracotomy
- Male
  Interventions: Other: Thoracotomy

INTERVENTIONS:
Other: Thoracotomy

SUMMARY:
Adequate analgesia in thoracic surgery is essential to prevent severe postoperative complications, especially respiratory problems. Current knowledge about gender-related differences in pain states generally more frequent and intense pain and more demand for analgesics in women. Results about postsurgical pain in particular are very inconclusive.

The investigators tried to find out if gender has an influence on postthoracotomy pain and analgesics requirement.

ELIGIBILITY:
Inclusion Criteria:

* open lung surgery between July 2010 and December 2014

Exclusion Criteria:

* redo-thoracotomy
* chest wall or rib resection
* other approach than lateral thoracotomy
* additional incision at other site (e.g. laparotomy)
* chest trauma
* mesothelioma
* hemofiltration or haemodialysis
* longer than one day stay at intensive care unit
* pre-existent chronic pain and/or chronic opioid intake
* short stay in hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2010-07-01; Primary Completion 2014-12-31 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scores | first 5 postoperative days
Analgesics requirement | first 5 postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Auinger, MD, Principal Investigator — Medical University of Graz; Freyja-Maria Smolle-Jüttner, Study Director — Medical University of Graz
Locations (1):
- Medical University of Graz, Division of Thoracic and Hyperbaric Surgery, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Auinger D, Sandner-Kiesling A, Striessnig A, Lindenmann J, Smolle J, Friedl H, Smolle-Juttner FM. Is There an Impact of Sex on Acute Postthoracotomy Pain? A Retrospective Analysis. Ann Thorac Surg. 2020 Apr;109(4):1104-1111. doi: 10.1016/j.athoracsur.2019.11.016. Epub 2019 Dec 28. PMID 31891695